CLINICAL TRIAL: NCT01396382
Title: Use of 68Ga-DOTATATE PET Scanning for Diagnosis and Treatment of Metastatic Neuroendocrine Tumors
Brief Title: 68Ga-DOTATATE PET Scan in Neuroendocrine Cancer
Acronym: 68Ga
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Ronald C. Walker MD, Professor of Clinical Radiology, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC GI 1136; 110588 (Other: Vanderbilt University Medical Center, Radiology Dept)
Record Dates: First submitted 2011-07-11; First posted 2011-07-18 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: Neuroendocrine Carcinoma
Keywords: neuroendocrine; neuroendocrine carcinoma; neuroendocrine tumor; carcinoid; carcinoid tumor; islet cell tumor; APUDoma; Gallium; PET Scan
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell; Apudoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-DOTATATE PET (Experimental): Patients will receive a 68Ga-DOTATATE PET scans
  Interventions: Radiation: 68Ga-DOTATATE PET scan

INTERVENTIONS:
Radiation: 68Ga-DOTATATE PET scan — 68Ga-DOTATATE will be given in tracer doses and injected intravenously to image tumors by Positron Emission Tomography (PET). Efficacy of the 68Ga-DOTATATE PET scan was assessed and compared to 111In-Pentetreotide scan and to scans with CT and/or MRI. Safety and toxicity were also assessed with pre-injection and post-imaging vital signs, pulse oximetry on room air, 12 lead ECGs, and blood laboratory tests, including tumor markers, liver and renal functions and blood counts, and direct patient questioning. Late delayed tumor markers, liver and renal functions and blood counts were assessed when available.

SUMMARY:
Neuroendocrine cancer is an unusual disease and often goes undetected by routine imaging. The 68Ga-DOTATATE PET scan is a new generation of scans that might have improved sensitivity and resolution specifically for neuroendocrine tumors. The investigators will scan people with this cancer and compare it to other conventional imaging methods to see if it improves patient care.

DETAILED DESCRIPTION:
Eligible participants will undergo baseline assessments at enrollment. Study participants will receive a one-time administration of 68GaDOTATATE and undergo a PET/CT imaging study. Scans will be performed with "negative" oral contrast (e.g. Volumen™ or equivalent), as many NETs involve the GI tract.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of neuroendocrine tumor
* At least 18 years of age
* Able to provide informed consent
* Karnofsky score greater than 50
* Females of childbearing potential must have a negative pregnancy test at screening/baseline

Exclusion Criteria:

* Serum creatinine >3.0 mg/dL (270 μM/L)
* Hepatic enzyme levels more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Use of any other investigational product or device within 30 days prior to dosing, or known requirement for any other investigational agent prior to completion of all scheduled study assessments.
* Patients with a body weight of 400 pounds or more or not able to enter the bore of the PET/CT scanner due to BMI, because of the compromise in image quality with CT, PET/CT and MRI that will result.
* Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.).
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Recognized concurrent active infection
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-03; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C. Walker, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Data are primarily imaging data and toxicity data submitted for peer-review publication and US FDA review, but not shared with a public data archive.

REFERENCES:
- [Result] Walker RC, Smith GT, Liu E, Moore B, Clanton J, Stabin M. Measured human dosimetry of 68Ga-DOTATATE. J Nucl Med. 2013 Jun;54(6):855-60. doi: 10.2967/jnumed.112.114165. Epub 2013 Mar 20. PMID 23516312
- [Result] Deppen SA, Liu E, Blume JD, Clanton J, Shi C, Jones-Jackson LB, Lakhani V, Baum RP, Berlin J, Smith GT, Graham M, Sandler MP, Delbeke D, Walker RC. Safety and Efficacy of 68Ga-DOTATATE PET/CT for Diagnosis, Staging, and Treatment Management of Neuroendocrine Tumors. J Nucl Med. 2016 May;57(5):708-14. doi: 10.2967/jnumed.115.163865. Epub 2016 Jan 14. PMID 26769865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This diagnostic study was conducted at Vanderbilt University/Ingram Cancer Center from March 2011-November 2013, at which time the study met target accrual and closed to accrual.
Pre-assignment Details: Ninety-nine patients were consented on this trial. Two consented patients were determined not eligible resulting in 97 patients on study.
Groups:
- 68Ga-DOTATATE PET Scan: 68Ga-DOTATATE PET scans performed on subjects. 68Ga-DOTATATE will be given in tracer doses and injected intravenously to image tumors by Positron Emission Tomography.
Period: Overall Study
Arm/Group | 68Ga-DOTATATE PET Scan
Started | 97
Completed | 97
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients with known or suspected pulmonary or gastroenteropancreatic (GEP) neuroendocrine tumors (NETS)
Groups:
- Imaging/Scans: 68Ga-DOTATATE PET scans performed on subjects. 68Ga-DOTATATE will be given in tracer doses and injected intravenously to image tumors by Positron Emission Tomography.
Arm/Group | Imaging/Scans
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (28.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 97

OUTCOME MEASURES:

1. Secondary Outcome: Number of Severe Adverse Events Occurences Resulting in Changes to Patient Treatment Plans, as a Measure of Safety and Tolerability
Description: Determine if any adverse effects are associated with the 68Ga-DOTATATE PET scan and the number of patients that experience them using NCI Common Terminology Criteria for Adverse Events v4.0, where: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening; Grade 5, death. Toxicities present at baseline and continuing without change in grade were excluded for assessment of this outcome measure.
Time Frame: at 1 year
Measure: Number; unit: participants
Groups:
- 68Ga-DOTATATE PET: 68Ga-DOTATATE PET scan will be administered to patients in tracer doses and injected intravenously to image tumors by Positron Emission Tomography.
Arm/Group | 68Ga-DOTATATE PET
Number analyzed (Participants) | 78
participants | 0

2. Primary Outcome: Number of Patients That Experienced a Change in Care Plans After 68GA-DOTATATE PET Scan
Description: Determine if the 68Ga-DOTATATE PET scan changes patient care plans compared to conventional imaging/diagnostic techniques (Octreoscan, MRI, CT, U/S).
Time Frame: at 1 year
Population: A major change in management is defined as:planned surgery cancelled, added, or a different type of surgery was planned, or a medication was added or stopped, or a new treatment modality (e.g. radiation) was added. A minor change was adjustment to planned surgery or radiation field, or in current medication dosage.
Measure: Number; unit: participants
Groups:
- 68Ga-DOTATATE PET: 68Ga-DOTATATE will be administered to patient in tracer doses and injected intravenously to image tumors by Positron Emission Tomography.
Arm/Group | 68Ga-DOTATATE PET
Number analyzed (Participants) | 78
participants
  Patients experienced a major change | 19
  Patients experienced a minor change | 9
  Patients experienced no change | 50

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 10 days minimum and up to 3 years, and/or until lost to follow-up. Some patients living outside the local region had limited long term follow-up.
Description: Toxicity data were compiled and individual patient test results pre-and-post-scans were compared. Non-systematic assessment was used for patients with limited long term follow-up.
Groups:
- 68Ga-DOTATATE PET Scan: Patients will receive 68Ga-DOTATATE PET scans. 68Ga-DOTATATE will be given in tracer doses and injected intravenously to image tumors by Positron Emission Tomography.
Arm/Group | 68Ga-DOTATATE PET Scan
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 51/97
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 68Ga-DOTATATE PET Scan (N=97)
hyperglycemia (Metabolism and nutrition disorders) | 11/62 (11)
hypertension (Vascular disorders) | 12 (12)
respiratory rate (Respiratory, thoracic and mediastinal disorders) | 6 (6)
white blood count (Investigations) | 5/75 (5)
Serum bilirubin mg/dl (Investigations) | 4/70 (4)
Serum alanine transaminase U/L (Investigations) | 7/70 (7)
Serum chloride mEg/L (Investigations) | 5/72 (5)
serum bicarbonate mEq/L (Investigations) | 8/67 (8)
Serum potassium (Metabolism and nutrition disorders) | 6/72 (6)

LIMITATIONS AND CAVEATS:
Long term follow-up of lab values was limited in some patients who lived outside the local region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes